CLINICAL TRIAL: NCT02227563
Title: tDCS & Auditory Hallucinations in Schizophrenia (AVH-SZ)
Brief Title: tDCS & Auditory Hallucinations in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants that fit inclusion criteria
Sponsor: Herzog Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Meiron 2013-3
Record Dates: First submitted 2014-05-20; First posted 2014-08-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
Keywords: dorsolateral prefrontal cortex; left superior temporal gyrus; auditory hallucinations; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Experimental): active tDCS
  Interventions: Device: Active tDCS
- control (Sham Comparator): sham (placebo) tDCS condition
  Interventions: Device: control

INTERVENTIONS:
Device: Active tDCS — repetitive daily tDCS sessions for a period of one week
  Arms: Active tDCS
Device: control
  Arms: control

SUMMARY:
The aim of this study is to evaluate tDCS effects on schizophrenia symptoms, particularly on auditory verbal hallucinations. tDCS applied with cathodal (inhibitory) electrode over the left temporal parietal junction and anodal (excitatory) electrode over the left dorsolateral prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* Primary diagnosis of Diagnostic and Statistical Manual, fifth edition, schizophrenia
* Persistent auditory verbal hallucinations
* Right handed
* Under stable doses of antipsychotic medication for ≥4 weeks
* Normal hearing by self-report and physical exam
* Use of effective method of birth control for women of childbearing capacity
* Capable to provide informed consent. For patients judged to be incapable to provide informed consent the legal guardian of the patient must agree to participation in the study and provide signed informed consent

Exclusion Criteria:

* Current or past history of substance dependence or abuse (excluding nicotine)
* Other current Axis I disorders
* History of seizure, epilepsy in self or first degree relatives, stoke, brain surgery, head injury, intracranial metal implants, known structural brain lesion, devices that may be affected by tDCS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Frequent and persistent migraines
* History of adverse reaction to neurostimulation
* Participation in study of investigational medication within 6 weeks
* Pregnancy
* Women who are breast-feeding
* Current significant laboratory abnormality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
change from baseline in auditory hallucination rating scale | 1 week post-treatment

SECONDARY OUTCOMES:
change in self-report quality of life scale from baseline | 1 week post treatment

OTHER OUTCOMES:
change from baseline in auditory event related potentials (ERP) | change in auditory ERP from baseline at 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Oded Meiron, PhD, Principal Investigator — Sarah Herzog Memorial Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel, Israel

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236